CLINICAL TRIAL: NCT06722118
Title: Corticoïdes Avant Extubation en réanimation pédiatrique : étude Multicentrique, Prospective, randomisée, Contre Placebo
Brief Title: Corticosteroids Before Extubation in Pediatric Intensive Care Unit
Acronym: COBEX-PED
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP220674
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Intensive Care Pediatric
Keywords: Corticosteroids; Intensive Care Pediatrics

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone IV
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone IV — IV-DXM 4mg/ml, injectable solution. Dosage of 0.25 mg/kg (maximum 5 mg per dose), prepared in a syringe of 5 to 10 ml and administered intravenously to the patient over 10 minutes every 6 hours. The treatment duration ranges from 6 hours (minimum of two doses: H0, H6) to 18 hours (maximum of four doses: H0, H6, H12, H18).
  Arms: Intravenous dexamethasone
Other: Placebo — Placebo: 0.9% NaCl solution, prepared in a syringe of 5 to 10 ml and administered intravenously to the patient over 10 minutes every 6 hours. The treatment duration ranges from 6 hours (minimum of two doses: H0, H6) to 18 hours (maximum of four doses: H0, H6, H12, H18).
  Arms: Placebo

SUMMARY:
Fifty to 60% of children admitted to a pediatric intensive care unit (PICU) are placed under invasive mechanical ventilation (MV) at least once during their stay. After extubation, about 30% of these patients will experience respiratory distress due to upper airway obstruction (RDUAO), and about one-third of these cases will require re-intubation. Treating this RDUAO extends the length of stay in the PICU.

Pre-extubation corticosteroid therapy has been validated in adults as a preventive treatment for the occurrence of RDUAO. However, the lack of robust data in pediatrics has not allowed for a consensus on the benefit of its use in children on MV in the PICU.

The investigators propose to conduct a randomized, multicenter, double-blind, placebo-controlled study evaluating the effect of intravenous dexamethasone (IV-DXM) before extubation on the incidence of RDUAO in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients intubated with an endotracheal tube with or without a cuff,
* Aged from 2 days post-term to 6 years,
* On mechanical ventilation for at least 36 hours,

And meeting the following extubation criteria:

* Extubation planned by the medical team
* Fraction of inspired oxygen (FiO2) ≤ 45%,
* Oxygen saturation measured by pulse oximeter ≥ 95% or appropriate according to the pathology,
* Positive end-expiratory pressure (PEEP) ≤ 8 cmH2O,
* Peak inspiratory pressure ≤ 22 cmH2O or presence of cough.
* Affiliated with a social security system,
* Collection of informed consent from the parental authority, by both parents or the legal guardian(s).

Exclusion Criteria:

* Refusal of consent by at least one parent or by the legal guardian(s),
* Patient with a contraindication to IV-DXM:

  * Uncontrolled local or general infection,
  * Active viral infections (hepatitis, herpes, chickenpox, shingles),
  * Live vaccines,
  * Severe coagulation disorders,
  * Ongoing gastrointestinal bleeding,
  * Known hypersensitivity to IV-DXM or one of its excipients.
* Patient participating in another interventional study involving human subjects or being in the exclusion period following a previous study involving human subjects, if applicable,
* Patient receiving State Medical Aid,
* Patient on long-term NIV,
* Known upper airway pathology (UAP) before intubation or at the time of extubation,
* History of UAP surgery within the month preceding inclusion,
* Any situation deemed incompatible with the child's participation in the trial at the discretion of the investigating physician,
* Decision to limit or stop therapeutic interventions.
* Premature patients aged less than 40 weeks of gestation
* Newborns aged less than 2 days after post-term birth

Ages: 2 Days to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 348 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of respiratory distress due to upper airway obstruction (RDUAO) | Within 48 hours post-extubation

SECONDARY OUTCOMES:
Cumulative incidence of reintubation due to RDUAO | Within 48 hours following a planned extubation
Odds ratios associated with the occurrence of RDUAO | Within 48 hours post-extubation
Number of days of hospitalization in pediatric intensive care unit (PICU) | Up to 28 days
Number of ventilator-free days in PICU | Up to 28 days
Number of days with non-invasive ventilation (NIV) post-extubation | Up to 28 days
Incidence of IV-DXM side effects | Up to 48 hours post-extubation

IPD SHARING:
Plan to Share IPD: Undecided